CLINICAL TRIAL: NCT02665780
Title: Assessing the Effect of Periodontal Debridement, Tongue Cleaning and Mouth Rinsing for the Treatment of Oral Malodour
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding was not secured
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Leeann Donnelly, Assistant Professor, Dept. Oral Biological and Medical Sciences, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H15-02159
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Halitosis
Keywords: halitosis, periodontal debridement, chemotherapeutics
MeSH Terms: conditions — Halitosis | interventions — Periodontal Debridement; Cetylpyridinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Periodontal debridement, tongue cleaning, mouth rinsing with 20ml Cetylpyridium Chloride daily for 24 weeks
  Interventions: Procedure: Periodontal debridement; Other: Cetylpyridium chloride

INTERVENTIONS:
Procedure: Periodontal debridement — teeth cleaning
Other: Cetylpyridium chloride — mouthrinse

SUMMARY:
This study evaluates the short and long term effect of dental cleaning and mouthrinsing for the treatment of bad breath

DETAILED DESCRIPTION:
The majority of bad breath producing bacteria can be found in pockets around the gums and the top of the tongue. It is generally agreed that one of the most effective means of controlling the production of bad breath gases from these bacteria is their mechanical removal. Tongue cleaning has shown consistent results in the reduction of bad breath, while dental cleaning has shown positive, but less conclusive results. The addition of a mouth rinse to mechanical measures has shown medium-term effectiveness, however there is currently no information available that describes the long-term impact of mechanical and chemical measures for the treatment of bad breath and the appropriate interval for follow-up and on-going management to prevent difficult cases.

ELIGIBILITY:
Inclusion Criteria:

Organoleptic score of 2 or more, and volatile sulfur compound score of greater than 1.5ng/10ml of hydrogen sulfide and 0.5ng/10ml of methyl mercaptan

-

Exclusion Criteria:

* Moderate to severe periodontal disease, systemic illness or dental disease associated with halitosis, antibiotic use in the past month, need for antibiotic prophylaxis for dental procedures and current smokers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Reduction of oral malodour below threshold | 1, 12, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Leeann Donnelly, PhD, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No